CLINICAL TRIAL: NCT00117819
Title: Dynamic SPECT Imaging With [123I] B-CIT in Individuals With Parkinsonian Syndrome (PS) and in Individuals at Risk for Parkinsonian Syndrome
Brief Title: A Study of Brain Imaging With Nuclear Medicine Technology in Individuals With and at Risk for Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Indiana University (Other); Albany Medical College (Other)
Responsible Party: Principal Investigator, Kenneth Marek, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: At-Risk
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Parkinsonian Syndrome
Keywords: parkinson; family history; diagnosis
MeSH Terms: conditions — Parkinsonian Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]ß CIT and SPECT imaging (Experimental): To assess [123I]ß-CIT and SPECT imaging
  Interventions: Drug: [123I]ß CIT and SPECT imaging

INTERVENTIONS:
Drug: [123I]ß CIT and SPECT imaging — To assess [123I]ß CIT and SPECT imaging
  Other Names: [123I]ß CIT; SPECT imaging

SUMMARY:
This study involves study participants who have been clinically diagnosed with parkinsonian syndrome or who are at-risk for parkinsonian syndrome, have a family history of parkinsonian syndrome or exposure to environmental toxins potentially associated with parkinsonian syndrome. Participants will have brain imaging to assess dopamine transporter density. The imaging data coupled with family history and environmental exposure data may provide important information about potential risk factors for parkinsonian syndrome.

DETAILED DESCRIPTION:
The brain imaging is conducted at the Institute for Neurodegenerative Disorders in New Haven, Connecticut. The imaging procedure occurs over a two day period.

On the first day participants are injected with [123I]ß CIT, an investigational radioactive material that localizes in the brain. Study participants will also have a thorough neurologic examination and standard neuropsychological testing, including testing of memory, concentration, abstraction and visual spatial functions.

Twenty-four hours later study participants return to the Institute for Neurodegenerative Disorders where an investigational scanning procedure will be used to obtain SPECT (single photon emission computed tomography) images of the brain.

Participants may be contacted to repeat these procedures every 12 to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 22 years or older
* A clinical diagnosis of Parkinson's disease (PD), positive family history of PD and/or potential exposure to environmental toxins
* Normal screening laboratory studies

Exclusion Criteria:

* Pregnancy
* Psychiatric disease other than history of depression
* Significant medical disease including abnormalities on screening

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2001-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
CIT uptake is the Specific: Nondisplaceable striatal uptake ratio | 2 yrs

SECONDARY OUTCOMES:
CIT uptake measures from at-risk individuals will be compared with healthy subjects. | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Marek, MD, Principal Investigator — President and Senior Scientist
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Koller WC, Langston JW, Hubble JP, Irwin I, Zack M, Golbe L, Forno L, Ellenberg J, Kurland L, Ruttenber AJ, et al. Does a long preclinical period occur in Parkinson's disease? Neurology. 1991 May;41(5 Suppl 2):8-13. No abstract available. PMID 2041599
- [Background] Marek, K., J. Seibyl, et al. (1999). "[123I] ß-CIT/SPECT: Assessment of determinants of variability in progression of Parkinson's disease." Neurology 52: A91-92.
- [Background] Marek, K., J. Seibyl, et al. (1996). "Dopamine transporter and receptor imaging in Parkinsonism. (Presented at the 4th International Congress of Movement Disorders, Vienna, Austria; June, 1996.)." Mov Dis 6.
- [Background] Morrish PK, Sawle GV, Brooks DJ. An [18F]dopa-PET and clinical study of the rate of progression in Parkinson's disease. Brain. 1996 Apr;119 ( Pt 2):585-91. doi: 10.1093/brain/119.2.585. PMID 8800950
- [Background] Seibyl JP, Marek KL, Quinlan D, Sheff K, Zoghbi S, Zea-Ponce Y, Baldwin RM, Fussell B, Smith EO, Charney DS, van Dyck C, et al. Decreased single-photon emission computed tomographic [123I]beta-CIT striatal uptake correlates with symptom severity in Parkinson's disease. Ann Neurol. 1995 Oct;38(4):589-98. doi: 10.1002/ana.410380407. PMID 7574455